CLINICAL TRIAL: NCT02513381
Title: The Effect of Colecalciferol (Vitamin D) on Hormonal, Metabolic and Cardiovascular Risk Factors in Patients With Polycystic Ovary Syndrome (PCOS) - a Double Blind Randomised Placebo-controlled Study
Brief Title: Effect of Vitamin D on Hormonal, Metabolic and Cardiovascular Risk Factors in Patients With Polycystic Ovary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hull University Teaching Hospitals NHS Trust (Other Government)
Collaborators: University of Hull (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 14/YH/1125
Record Dates: First submitted 2015-07-23; First posted 2015-07-31 (Estimated); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Vitamin D3, 3200IU (Active Comparator): Each participant will receive either Vitamin D3, 3200IU or Placebo daily for three months.
  Interventions: Other: Vitamin D3, 3200IU
- Placebo (Placebo Comparator): Each participant will receive either Vitamin D3, 3200IU or Placebo daily for three months.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Vitamin D3, 3200IU — Each participant will receive either Vitamin D3, 3200IU or Placebo daily for three months.
  Arms: Vitamin D3, 3200IU
Other: Placebo — Each participant will receive either Vitamin D3, 3200IU or Placebo daily for three months.
  Arms: Placebo

SUMMARY:
This is a double blind randomised placebo-controlled study involving women with polycystic ovary syndrome (PCOS). The patients will be randomised either to Vitamin D 3200 IU or placebo for three months. The main hypothesis of this study is "Vitamin D improves hormonal, metabolic and cardiovascular risk markers in women with PCOS".

DETAILED DESCRIPTION:
Polycystic ovary syndrome (PCOS) is a very common condition in women which could present with irregular periods, excessive hair growth on body, acne and cysts in the ovaries. PCOS is also associated with increased risk of problems later in life like diabetes, high cholesterol levels and heart disease. One of the risk factors for having increased incidence of such problems in PCOS patients could be low vitamin D levels as many women with polycystic ovary syndrome (PCOS) are vitamin D deficient. Vitamin D supplementation may have a beneficial effect on insulin levels and fat around the abdomen. It has been seen in previous research studies that low level of vitamin D is related to a greater risk of diabetes and heart disease. Low vitamin D levels are also associated with fat in the liver. The amount of fat in the liver is a sign of early liver disease. So, in this study the investigators want to supplement women having PCOS and vitamin D deficiency with vitamin D (3,200 IU) and examine the effects on hormones related to PCOS and risk factors for diabetes and heart disease in them.

ELIGIBILITY:
Inclusion Criteria:

1. Caucasian women, aged 18-45 years, with confirmed diagnosis of PCOS based on all three diagnostic criteria of the Rotterdam consensus [21].
2. Irregular periods with raised FAI
3. Vitamin D < 50 nmol/L.

Exclusion Criteria:

1. Non-classical 21-hydroxylase deficiency, hyperprolactinaemia, Cushing's disease and androgen-secreting tumours will be excluded by appropriate tests if clinically indicated.
2. Any concurrent illness including type 2 diabetes, subjects who are on any medication (including medications that interfere with calceotrophic hormones) for the preceding 6 months.
3. Women planning to conceive.
4. Women who are using any oral or implantable contraceptives or any other treatments likely to affect ovarian function, insulin sensitivity or lipids for at least 3 months before entering the study. Stable dose of metformin for 3 months is allowed. Subjects will be advised to use barrier contraception during the study period.
5. eGFR<60.
6. Hypersensitivity to vitamin D or any of the excipients in the product.
7. Peanut or soya allergy.
8. Nephrolithiasis.
9. Diseases or conditions resulting in hypercalcaemia and/or hypercalciuria.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2015-07; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Cardiovascular risk assessment by hs-CRP, HOMA (fasting glucose & insulin) and fasting lipid profile | Three months supplementation with Vitamin D3 3200IU or placebo

SECONDARY OUTCOMES:
Hormonal parameters including testosterone, SHBG and FAI. | Three months supplementation with Vitamin D3 3200IU or placebo
Inflammatory marker hs-CRP | Three months supplementation with Vitamin D3 3200IU or placebo
Endothelial function by EndoPAT | Three months supplementation with Vitamin D3 3200IU or placebo

CONTACTS AND LOCATIONS:
Overall Officials: Thozhukat Sathyapalan, MD, FRCP, Principal Investigator — University of Hull
Locations (1):
- Michael White Centre for Diabetes and Endocrinology, Hull, East Yorkshire, United Kingdom

REFERENCES:
- [Result] Javed Z, Papageorgiou M, Deshmukh H, Kilpatrick ES, Mann V, Corless L, Abouda G, Rigby AS, Atkin SL, Sathyapalan T. A Randomized, Controlled Trial of Vitamin D Supplementation on Cardiovascular Risk Factors, Hormones, and Liver Markers in Women with Polycystic Ovary Syndrome. Nutrients. 2019 Jan 17;11(1):188. doi: 10.3390/nu11010188. PMID 30658483